CLINICAL TRIAL: NCT06347081
Title: Efficacy of a Long-Pulsed 1064 nm Nd:YAG Laser (Neodymium-doped Yttrium Aluminium Garnet) for Hypertrophic Scars: A Randomized Controlled Trial
Brief Title: Effect of Nd-YAG Laser on Hypertrophic Scar
Acronym: Nd-YAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noha F. mahmoud, Assis prof of rehabilitation, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/00449
Record Dates: First submitted 2024-03-27; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Hypertrophic Scar
Keywords: Nd-YAG laser
MeSH Terms: conditions — Cicatrix, Hypertrophic

STUDY DESIGN:
Intervention Model Description: one treatment one control group
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Patients received standard medical care, nursing, physiotherapy, and a sham laser during the course of treatment
  Interventions: Procedure: Nd- YAG laser at 532nm wavelength
- Laser group (Active Comparator): Patients received 532 nm laser radiation in addition to standard medical care, nursing, and physiotherapy.
  Interventions: Procedure: Nd- YAG laser at 532nm wavelength

INTERVENTIONS:
Procedure: Nd- YAG laser at 532nm wavelength — Nd-YAG laser at 532nm wavelength every 2 weeks for 14 sessions. patients will also receive standard medical care, nursing, physiotherapy

SUMMARY:
A hypertrophic scar is a serious health concern in the industrialized world. Two groups of patients were treated with standard medical care. The experimental group received additional laser therapy. scar assessment was measured immediately before treatment, after 3, and 7 months.

T test for comparison before-treatment between the control and study groups. ANOVA with repeated measures test for comparison among other measures.

DETAILED DESCRIPTION:
Background: A hypertrophic scar is a serious health concern in the industrialized world. Objective: The impact of this study was to investigate the effect of the Nd-YAG laser at 532nm wavelength on hypertrophic scars. Patients and methods: Forty male and female patients with hypertrophic scars, ranging in age from fifteen to forty-five, were recruited from the burn patients' clinic within the Faculty of Physical Therapy, Cairo University, for this study. They were randomized into two equivalent groups. Group A (the control group) consisted of 20 patients who were given standard medical care, nursing, physiotherapy, and a sham laser during the course of treatment. In contrast, Group B (the study group) consisted of 20 patients who were given 532 nm laser radiation in addition to standard medical care, nursing, and physiotherapy. Treatment was conducted every 2 weeks for 14 sessions. Outcome measures included Vancouver Scar Scale score and scar volume. The assessment procedures were applied before the initiation of treatment (Pre), after 3 months (Post1) and after 7 months (Post 2) from the beginning of the treatment.

ELIGIBILITY:
IInclusion Criteria:

• Adult patients with hypertrophic scars.

Exclusion Criteria:

* Patients were excluded if they had taken oral retinoids in the last year.
* Patients had any skin defects.
* Patients had any history of photosensitivity.
* Patients experienced active skin diseases in the treatment regions (such as psoriasis, cancer, or autoimmune disease).

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
hypertrophic scar maturation | before treatment,12 weeks, and then 28 weeks of the treatment.
  Changes in the scars' color, vascularity, elevation, and pliability were evaluated and scored using the Vancouver scale (VSS). VSS is from 0 to 14. A lower value indicates a better scar.
hypertrophic scar volume | before treatment,12 weeks, and then 28 weeks of the treatment.
  Scar volume was determined using the negative-positive moulage method.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo, Egypt